CLINICAL TRIAL: NCT03413267
Title: Impact of Food Structure on Micronutrient Biovailability in Human
Brief Title: Impact of Food Structure on Micronutrient Bioavailability in Human
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Françoise Nau (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government); University Hospital, Clermont-Ferrand (Other); Université d'Auvergne (Other)
Responsible Party: Sponsor-Investigator, Françoise Nau, PhD, Professor, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Organization: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MicroNut; 2017-A01996-47 (Other: French Health Agency)
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Food Structure Impact on Micronutrient Bioavailability
Keywords: micronutrient; bioavailability; bioaccessibility; food structure; food texture
MeSH Terms: interventions — BAG 0177

STUDY DESIGN:
Intervention Model Description: Bioavailability protocol : each volunteer participates in 4 interventions (4 food matrices), during 4 different days (one food matrix per day). At least 3 weeks between each intervention day. An intervention consists in food matrix ingestion (t=0) and blood sampling for 8 h postprandial (10 sampling times).
  Mastication protocol : each volunteer participates in 1 session during which 2 solid matrices will be studied. For each matrix, 13 samples are proposed to the volunteer; food bolus are collected just before the volunteer feels the need of swallowing.
Masking Description: Because the food matrices ingested by the volunteers have different aspects, no masking is really possible. However, blood samples will be analyzed by partners without knowledge of the matrix that has been ingested.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Custard (Experimental): The food matrix ingested (once by each volunteer) is a custard containing 1250µg vitamin D (=50 000 UI), 12µg vitamin B12, 1000µg vitamin B9 and 20 mg lutein
  Interventions: Other: Custard
- Flan (Experimental): The food matrix ingested (once by each volunteer) is a flan containing 1250µg vitamin D (=50 000 UI), 12µg vitamin B12, 1000µg vitamin B9 and 20 mg lutein
  Interventions: Other: Flan
- Sponge cake (Experimental): The food matrix ingested (once by each volunteer) is a sponge cake containing 1250µg vitamin D (=50 000 UI), 12µg vitamin B12, 1000µg vitamin B9 and 20 mg lutein
  Interventions: Other: Sponge cake
- Biscuit (Experimental): The food matrix ingested (once by each volunteer) is biscuits containing 1250µg vitamin D (=50 000 UI), 12µg vitamin B12, 1000µg vitamin B9 and 20 mg lutein
  Interventions: Other: Biscuit

INTERVENTIONS:
Other: Custard — Food matrix: custard (liquid emulsion)
  Arms: Custard
Other: Flan — Food matrix: flan (soft gel)
  Arms: Flan
Other: Sponge cake — Food matrix: sponge cake (porous and spongy)
  Arms: Sponge cake
Other: Biscuit — Food matrix: biscuit (thick and crunchy)
  Arms: Biscuit

SUMMARY:
The nutritional quality of foods strongly depends on the structure / texture of foods, because of the impact on food disintegration, and then on digestion process and nutrient utilization by the human body. However, this relationship between food structure and nutrient bioavailability is still widely unknown.

MicroNut project aims at demonstrating and evaluating in humans the impact of structure / texture changes on micronutrient bioavailability. In order to do this, four complex food matrices, with constant composition but different structures / textures, and as close as possible to real foods have been designed and are evaluated in the present study. A mixture of egg and plant proteins is the basis of these lipoprotein matrices in which four micronutrients will be followed up : two lipophilic (vitamin D and lutein) and 2 hydrophilic (vitamins B9 and B12).

DETAILED DESCRIPTION:
The main objective consists in understanding how food structure / texture impacts on micronutrient bioavailability. The second objective consists in studying food disintegration at oral phase (in the mouth) and the consequences on the bioaccessibility of hydrophilic vitamins in saliva.

The clinical study is open, monocentric, controled and randomized, in a cross experimental design.

The included volunteers (n=12) will participate in the whole two protocols. The first protocol is related to the study of vitamins B9, B12, D and lutein bioavailability during 8h kinetics, after ingestion of a food matrix (custard, biscuit, flan or sponge cake). The second protocol is related to the study of hydrophilic vitamin release during mastication of two of these matrices (biscuit and sponge cake).

The study is not performed in a double blind way. However, the measure bias will be limited because of the standardized and objective characteristic of the main criteria. Moreover, biological samples will be analysed by the same partners of the project. Each subject will be his own control, so that confusion factors related to individual variability will be eliminated.

The monocentric characteristic of the study, the low number of subjects and the expertise of the involved staff will enable to limit the number of missing data.

The randomization (latin square) has been established by a bio-statistician of the project before the study started. A document describing the randomization proceeding is confidentially kept.

ELIGIBILITY:
Inclusion Criteria:

* no smoking since 6 months at least
* no pathology and no medical treatment
* no history of calcium lithiasis
* BMI >=20 and <=30 kg/m²
* normal biological status
* no dislike for the food tested
* good dental health, no pain, no treatment in progress, no orthodontics since 3 years

Exclusion Criteria:

* hypercalcemia (>2.52 mmol/L), hyperphosphoremia (>1.58 mmol/L)
* known pathology
* allergy or intolerance to one of the food matrix components (egg, vitamins B12, B9, D, lutein, pea, gluten)
* intake of food supplements and/or UVdose for the 3 months before the study, except enriched foods
* exposure to UV during the 2 weeks before the study and all along the study
* vitamin D < 80µg/L

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2018-04-19 (Actual); Study Completion 2018-04-19 (Actual)

PRIMARY OUTCOMES:
Quantitative analysis of vitamin D, B9, B12 and lutein in blood | 8 hours
  Blood sampling before (T-30min to determine basal concentrations) and after food matrix ingestion (T0) for 8 h postprandial (10 sampling between 30 and 480min postprandial) for vitamin D, B9, B12 and lutein measurement in plasma; vitamin D and lutein will be quantified by HPLC-DAD in the chylomicron fraction; vitamin B9 and B12 will be quantified by ELISA method
Quantitative analysis of vitamin B9 and B12 in the liquid fraction of food boluses and characterization of these boluses | one and half hour
  Normal mastication of food matrix and splitting out for characterization of food bolus: granulometry, rheology and vitamin B9 and B12 release in the liquid fraction (saliva + food water + rinsing water); each volunteer successively masticates 13 samples of each solid food matrix (biscuit and sponge cake); vitamin B9 and B12 will be quantified by ELISA method

CONTACTS AND LOCATIONS:
Overall Officials: Ruddy Richard, Prof, Principal Investigator — Centre de Recherche en Nutrition Humaine d'Auvergne
Locations (1):
- Centre de Recherche en Nutrition HUmaine d'Auvergne, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data for all outcome measures will be made available, only after joined consent of promotor and investigator. Data use and transfer to a third party will be performed according to the agreement signed as part of the grant funded by Qualiment